CLINICAL TRIAL: NCT00103324
Title: Phase II Study of GW572016 (NSC-727989) as First Line Therapy in Patients With Advanced or Metastatic Gastric Cancer
Brief Title: S0413 Lapatinib in Treating Patients With Locally Advanced or Metastatic Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03180; S0413; U01CA32102 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000409575 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage III Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well lapatinib works in treating patients with locally advanced or metastatic stomach cancer. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the confirmed response (complete and partial) probability in patients with advanced/metastatic gastric cancer treated with GW572016.

II. To assess the time to treatment failure and overall survival in this group of patients.

III. To assess the qualitative and quantitative toxicities associated with this regimen.

IV. To assess, in a preliminary manner, the relationship of protein expression and gene expression of EGFR, HER2 and markers of angiogenesis with clinical outcomes in patients treated with GW572016.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically or pathologically verified diagnosis of gastric cancer; patients must have locally advanced or distant metastatic disease (either recurrent or at primary diagnosis) that is not surgically curable

  * The pathologic confirmation of gastric cancer may be made from the metastatic site; biopsy of the primary tumor is not necessary; patients with pathologic confirmation of cancer from a metastatic site, along with clinical documentation of gastric involvement and no evidence of another primary are also eligible
  * Eligible pathologic type: patients may have any histological subtype including adenocarcinoma NOS, papillary carcinoma, adenocarcinoma, intestinal type, clear cell adenocarcinoma, mucinous carcinoma, signet ring cell carcinoma, undifferentiated carcinoma, carcinoma NOS; patients must not have carcinoid tumors or sarcomas
* Patients must have measurable disease; x-rays, scans, or physical examinations for measurable disease must have been completed within 28 days prior to registration; x-rays, scans or physical examinations for non-measurable disease must have been completed within 42 days prior to registration,; all disease must be assessed
* Patients must be willing to have specimens submitted; the paraffin embedded specimens must be available for submission
* Patients may have had prior surgery for their gastric cancer; patients must be at least 2 weeks beyond surgery, and recovered from all effects of surgery
* Patients may have received prior chemotherapy, hormonal therapy, immunotherapy, radiation or chemoradiotherapy as neoadjuvant or adjuvant treatment but this must have been completed at least 6 months prior to documented recurrence or metastatic disease; patients must not have received previous treatment for metastatic disease

  * If patient received radiation therapy, the site of measurable disease must be outside of the radiation field
* Patients must not have had prior therapy with EGFR targeting therapies
* Patients must have a Zubrod performance status of 0-1
* Leukocytes >= 3,000/mcl
* Platelets >= 100,000/mcl
* AGC >= 1,500/mcl
* Serum transaminase (SGOT or SGPT) =< 2.5 x IULN; patients with liver metastases must have SGOT/SGPT =< 5 x IULN
* Bilirubin =< IULN
* Serum creatinine =< IULN OR measured creatinine clearance > 60 mL/min OR estimated creatinine clearance> 60 mL/min
* Patients must have cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan; note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution
* Patients must either be able to swallow and/or receive enteral medications via gastrostomy feeding tube; patients with intractable nausea or vomiting are not eligible; patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis) are not eligible
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016
* There must be no plans for the patient to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of their cancer while on this protocol
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with GW572016
* Pregnant or nursing women are not eligible because of the risk of fetal harm; nursing women may participate only if nursing is discontinued, due to the possibility of harm to nursing infants from this treatment regimen; women/men of reproductive potential must have agreed to use an effective contraceptive method
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in remission or any other cancer from which the patient has been disease-free for 5 years
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day

  * In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Statistical Center in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Confirmed response probability (complete and partial) | Up to 2 years

SECONDARY OUTCOMES:
Time to treatment failure | From the date of registration to the date of first observation of progressive disease, death due to any cause, symptomatic deterioration, or early discontinuation of treatment, assessed up to 2 years
Overall survival | From date of registration to date of death due to any cause, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States